CLINICAL TRIAL: NCT03656471
Title: Comparison of Subjective Experiences Between Patients Receiving Clear Aligners or Fixed Appliances During the Initial Stage of Orthodontic Treatment
Brief Title: Comparison of Subjective Experiences Between Patients Receiving Clear Aligners or Fixed Appliances
Status: Completed | Type: Observational
Sponsor: West China Hospital (Other)
Responsible Party: Principal Investigator, Meiya Gao, Principal Investigator, West China Hospital
Other Study IDs: WCHSIRB-D-2013-108
Record Dates: First submitted 2018-08-30; First posted 2018-09-04 (Actual); Last update posted 2018-09-04 (Actual); Status verified 2018-08

CONDITIONS: Pain; Anxiety; Quality of Life
MeSH Terms: conditions — Pain; Anxiety Disorders | interventions — Orthodontic Appliances, Fixed

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 14 Days
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Clear aligner group: Patients receiving clear aligner treatments for their malocclusions
  Interventions: Device: clear aligners or fixed appliances
- Fixed appliance group: Patients receiving fixed appliance treatments for their malocclusions
  Interventions: Device: clear aligners or fixed appliances

INTERVENTIONS:
Device: clear aligners or fixed appliances — Patients choose clear aligners or fixed appliances to treat their malocclusions

SUMMARY:
This study aimed to compare experiences between adult patients receiving clear aligners and fixed appliances during the initial stage of orthodontic treatments.

DETAILED DESCRIPTION:
Patients receiving either clear aligner treatments were enrolled in this study. During the same time period, patients receiving fixed orthodontic treatments well-matched with clear-aligner patients by similar ages (difference < 3 years), same gender and similar levels of severity of malocclusion [similar Index of Complexity Outcome and Need (ICON) level] were enrolled.The two groups were well-matched with ages, gender and levels of malocclusion severity. Pain perception, anxiety and quality of life were assessed through visual analogue scale (VAS), state-trait anxiety inventory (STAI) and oral health impact profile-14 (OHIP-14), respectively.

ELIGIBILITY:
Inclusion Criteria:

* Must be 18 years of age or older;
* Must be in good general health;
* Upper and lower arches were both involved in two groups;
* The fixed appliances group must be treated with wires and brackets only with the initial arch wire of 0.012 NiTi ;
* Must be willing to sign and give written informed consent in accordance with institutional and federal guidelines.

Exclusion Criteria:

* Once been undergoing with orthodontic treatment;
* Experienced tooth ache recently;
* Been diagnosed with contagious and/or systematical diseases;
* Have taken any kind of painkillers three days before the initial treatment;
* When Trait Anxiety Inventory (T-AI) shows a score believed to define a psychological state of over anxiety (male over 53 points and female over 55 points).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients receiving either clear aligner or conventional fixed appliance treatments from December 2013 to December 2015 in West China Hospital of Stomatology were enrolled in this study.
Sampling Method: Non-Probability Sample
Enrollment: 160 (Actual)
Dates: Start 2013-12-03 (Actual); Primary Completion 2015-12-03 (Actual); Study Completion 2016-02-01 (Actual)

PRIMARY OUTCOMES:
The chronological changes in pain perception | Baseline, Day 1, Day 2，Day 3，Day 4，Day 5，Day 6，Day 7,and Day 14
  The chronological changes in pain perception during the fortnight of orthodontic treatment were assessed through visual analogue scale (VAS). Participant is asked to place a line perpendicular to the VAS line.The score is determined by measuring the distance (mm) on the 10-cm line between the "no pain"anchor and the patients' mask,providing a range of scores from 0-100. A higher score indicates greater pain.

SECONDARY OUTCOMES:
The chronological changes of anxiety level | Baseline, Day 1,Day 3,Day 5,Day 7 and Day 14
  Secondary outcomes concerning chronological changes of anxiety were assessed before and after orthodontic treatments through state-trait anxiety inventory (ST-AI). A higher score indicates higher anxiety level.
The chronological changes in quality of life | Baseline,Day 1 ,Day 7 and Day 14
  Secondary outcomes concerning chronological changes of anxiety of life were assessed before and after orthodontic treatments through oral health impact profile-14 (OHIP-14).A higher score indicates lower quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Hu Long, PhD, Principal Investigator — West China Hospital of Stomatology, Sichuan University, Chengdu, China